CLINICAL TRIAL: NCT04832880
Title: Factorial, Multicentric, Randomized Clinical Trial of Remdesivir and Immunotherapy in Combination With Dexamethasone for Moderate COVID-19 (the AMMURAVID Trial)
Brief Title: Factorial Randomized Trial of Rendesivir and Baricitinib Plus Dexamethasone for COVID-19 (the AMMURAVID Trial)
Acronym: AMMURAVID
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Enrico Tombetti, Assistant Professor, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The AMMURAVID trial; 2020-001854-23 (EudraCT Number)
Record Dates: First submitted 2020-10-12; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: remdesivir; baricitinib; dexamethasone
MeSH Terms: conditions — COVID-19 | interventions — baricitinib; remdesivir; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Factorial design with four-stages (K=4). Three interim analyses are pre-planned. At each stage, the use of remdesivir and/or baricitinib might be suspended due to futility or ef-ficacy. Overall, we will accept a two-sided alpha error of alpha=0.05 and a beta error of β=0.10.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control arm (dexamethasone arm) (Experimental): IV dexamethasone 6 mg for 10 days
  Interventions: Drug: Dexamethasone
- Remdesivir arm (Experimental): IV dexamethasone 6 mg for 10 days + remdesivir IV 200 mg on day 1, followed by 100 mg die until day 10
  Interventions: Drug: Remdesivir; Drug: Dexamethasone
- Baricitinib arm (Experimental): IV dexamethasone 6 mg for 10 days + baricitinib 4 mg die for 10 days. For patients aged > 75 years or estimated GFR < 60 ml/min*1.73m2, baricitinib dose is reduced to 2 mg for 10 days.
  Interventions: Drug: Baricitinib Oral Tablet [Olumiant]; Drug: Dexamethasone
- Remdesivir + baricitinib arm (Experimental): IV dexamethasone 6 mg for 10 days + remdesivir IV 200 mg on day 1, followed by 100 mg die until day 10 + baricitinib 4 mg die for 10 days.
  For patients aged > 75 years or estimated GFR < 60 ml/min*1.73m2, baricitinib dose is reduced to 2 mg for 10 days.
  Interventions: Drug: Baricitinib Oral Tablet [Olumiant]; Drug: Remdesivir; Drug: Dexamethasone

INTERVENTIONS:
Drug: Baricitinib Oral Tablet [Olumiant] — Baricitinib 4 mg die (2 mg for patients aged > 75 years) for 10 days.
  Other Names: Olumiant
  Arms: Baricitinib arm; Remdesivir + baricitinib arm
Drug: Remdesivir — Intravenous remdesivir 200 mg on day 1, followed by remdesivir 100 mg die until day 10
  Other Names: Veklury
  Arms: Remdesivir + baricitinib arm; Remdesivir arm
Drug: Dexamethasone — Intravenous dexamethasone 6 mg for 10 days

SUMMARY:
Background:

In the current worldwide medical emergency, a rapid identification of effective therapeutic strategy is crucial. So far, therapy with dexamethasone, remdesivir and baricitinib have been associated with evidence of impact on the clinical impact on COVID-19, but the effect of baricitinib and remdesivir in combination with dexamethasone.

The AAMMURAVID trial is endorced and supported by the Italian Regulatory agency (AIFA-Agenzia Italiana del Farmaco)

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 18 years able to provide a valid informed consent to the study
* Documented COVID-19 by direct testing (positive PCR), with lung infiltrates at imaging (Chest-X ray or CT) and requirement of oxygen supplementation
* Less than 10 days form symptoms onset
* Cytokine storm, using the criteria developed at Temple University (all of the three below criteria):

  * CRP > 46 mg/l
  * Ferritin > 250 ng/ml
  * One variable of each of the three clusters below

    * Cluster 1

      * Albumin < 2.8 g/dl
      * Lymphocytes <10.2 % of WBC
      * Absolute neutrophil count > 11400/mm3
    * Cluster 2

      * ALT > 60 U/L
      * AST > 87 U/L
      * D-dimers > 4930 µg/l fibrinogen-equivalent-units (FEU).
      * LDH >416 U/L
      * High sensitivity troponin > 1.09 ng/ml
    * Cluster 3

      * Anion Gap at arterial blood gas < 6.8 mM
      * Chloride > 106 mM
      * Potassium > 4.9 mM
      * BUN:creatinine ratio > 29
* PaO2/FiO2 200-400 mmHg, while in oxygen therapy or continuous positive airway pressure (C-PAP)
* For women of childbearing potential and men: agreement to use contraception in the case of heterosexual intercourses before day 28 with a failure rate < 1% per year (bilateral tubal ligation, male sterilisation, hormonal contraceptives inhibiting ovulation, hormone-release or copper intrauterine devices). For men enrolled in the study, condom use is allowed.

Exclusion criteria:

* Orotracheal intubation or ECMO support
* Active solid / hematologic cancer (including invasive non-melanoma skin cancer)
* Hypersensitivity or contra-indications to one of the investigational agents (including history of deep vein thrombosis / pulmonary thromboembolism within 12 weeks prior to screening)
* Other active concurrent viral, fungal or bacterial infections (including active tuberculosis/latent TB treated for less than 4 weeks, HIV and HCV/HBV infections)
* Pregnancy/breastfeeding
* Incapability to provide a valid informed consent (including age < 18 years old)
* Heart failure with NYHA >= 2 or any acute cardiac or vascular event requiring therapy in the previous 12 months
* Chronic renal failure (baseline GFR < 45 ml/min*1.73m2)
* Liver cirrhosis moderate / severe (Child-Pugh B or C)
* Chronic respiratory failure requiring O2 therapy or ventilation therapy at home
* Blood neutrophils <1000/mcL, platelet <50000/mcL, Hb levels <80 g/l
* ALT/AST > 5 times UNL
* Use of any biologic agent or small molecule inhibitor and other investigational drugs in the previous 4 weeks or 5 half-lives (whichever is longer). Specific cut-offs for wash-out are required for the following therapies:

  * B-cell targeted therapies: 24 weeks or 5 half-lives (whichever is longer)
  * TNF-inhibitors: 2 weeks or 5 half-lives (whichever is longer)
  * JAK-inhibitors: 1 week or 5 half-lives (whichever is longer)
* Use of other immunosuppressive agents in the last 3 months (chronic use of topical steroids and systemic steroids with a dose ≤5 mg of prednisone equivalents is allowed)
* Use of any other investigational therapy for COVID-19 (including IV immunoglobulins, convalescent COVID-19 plasma or monoclonal antibodies)
* Impossibility to discontinue Strong inhibitors of OAT3 (such as probenecid) at study entry
* Any other condition judged by the local investigator as a contra-indication to eligibility
* Subjects who have received live vaccines within 4 weeks before the study or are planned to receive live vaccine in the first months after study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2021-04-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of very severe respiratory failure or mortality | Day1-Day 28
  Composite outcome: Development of very severe respiratory failure (PaO2/FiO2 <150 mmHg) or mortality

SECONDARY OUTCOMES:
Prevention of mortality | Day 7
  Proportion of dead patients
Prevention of mortality | Day 14
  Proportion of dead patients
Prevention of mortality | Day 21
  Proportion of dead patients
Prevention of mortality | Day 28
  Proportion of dead patients
Prevention of mortality | Day 1-28
  Survival analysis
Prevention of very severe respiratory failure | Day 7
  Proportion of patients with PaO2/FiO2 <150 mmHg
Prevention of very severe respiratory failure | Day 14
  Proportion of patients with PaO2/FiO2 <150 mmHg
Prevention of very severe respiratory failure | Day 21
  Proportion of patients with PaO2/FiO2 <150 mmHg
Prevention of very severe respiratory failure | Day 28
  Proportion of patients with PaO2/FiO2 <150 mmHg
Prevention of very severe respiratory failure | Day 1-28
  Time to development very severe respiratory failure (PaO2/FiO2 <150 mmHg)
Prevention of very severe respiratory failure or mortality | Day 7
  Composite outcome: Development of very severe respiratory failure (PaO2/FiO2 <150 mmHg) or mortality
Prevention of very severe respiratory failure or mortality | Day 14
  Composite outcome: Development of very severe respiratory failure (PaO2/FiO2 <150 mmHg) or mortality
Prevention of very severe respiratory failure or mortality | Day 21
  Composite outcome: Development of very severe respiratory failure (PaO2/FiO2 <150 mmHg) or mortality
Incidence of Adeverse Events | Day 7
  Proportion of number of AEs and SAEs (according to the Common Terminology Criteria for Adverse Events -CTCAE, Version 5.0)
Incidence of Adeverse Events | Day 14
  Proportion of number of AEs and SAEs (according to the Common Terminology Criteria for Adverse Events -CTCAE, Version 5.0)
Incidence of Adeverse Events | Day 21
  Proportion of number of AEs and SAEs (according to the Common Terminology Criteria for Adverse Events -CTCAE, Version 5.0)
Incidence of Adeverse Events | Day 28
  Proportion of number of AEs and SAEs (according to the Common Terminology Criteria for Adverse Events -CTCAE, Version 5.0)
Incidence of bacterial/fungal infections | Day 7
  Rate of bacterial/fungal infections
Incidence of bacterial/fungal infections | Day 14
  Rate of bacterial/fungal infections
Incidence of bacterial/fungal infections | Day 21
  Rate of bacterial/fungal infections
Incidence of bacterial/fungal infections | Day 28
  Rate of bacterial/fungal infections
Reduction of the requirements of orotracheal intubation/ECMO | Day 7
  Proportion of patients requiring orotracheal intubation/ECMO
Reduction of the requirements of orotracheal intubation/ECMO | Day 14
  Proportion of patients requiring orotracheal intubation/ECMO
Reduction of the requirements of orotracheal intubation/ECMO | Day 21
  Proportion of patients requiring orotracheal intubation/ECMO
Reduction of the requirements of orotracheal intubation/ECMO | Day 28
  Proportion of patients requiring orotracheal intubation/ECMO
Reduction of the requirements of orotracheal intubation/ECMO | Day 1-28
  Days with orotracheal intubation/ECMO
Evolution of the NEWS-2 score | Day 1-28
  Course in the National Early Warning Score-2 score (0-20, with higher scores worse)
Evolution of the MELD score | Day 1-28
  Course in the Model for End-Stage Liver Disease score (scores >=6, higher scores worse)
Velocity in clinical improvement | Day 1-28
  Time to clinical improvement (defined as one of the following: a) discharge, b) absent ventilator support with NEWS-2 score ≤3 and MELD ≤13)
Velocity in discharge | Day 1-28
  Time to discharge
Velocity in discharge | Day 7
  Proportion of discherged patients
Velocity in discharge | Day 14
  Proportion of discherged patients
Velocity in discharge | Day 21
  Proportion of discherged patients
Velocity in discharge | Day 28
  Proportion of discherged patients
Fever disappearance | Day 7
  Proportion of patients on persistent defervescence (last day of T<37.0°C, without recurrent T>37.0° for at least 4 days)
Fever disappearance | Day 14
  Proportion of patients on persistent defervescence (last day of T<37.0°C, without recurrent T>37.0° for at least 4 days)
Fever disappearance | Day 21
  Proportion of patients on persistent defervescence (last day of T<37.0°C, without recurrent T>37.0° for at least 4 days)
Fever disappearance | Day 28
  Proportion of patients on persistent defervescence (last day of T<37.0°C, without recurrent T>37.0° for at least 4 days)
Fever disappearance | Day 1-28
  Time to persistent defervescence persistent defervescence (last day of T<37.0°C, without recurrent T>37.0° for at least 4 days)
Changes in periperal blood leukocyte number | Day 1-28
  Course of periperal blood leukocyte number
Changes in periperal blood neutrophils counts | Day 1-28
  Comparison of the course of neutrophils counts at full blood counts among the treatment arm, as assessed by repeated measures analysis.
Changes in periperal blood lymphocytes | Day 1-28
  Comparison of the course of lymphocytes counts at full blood counts among the treatment arm, as assessed by repeated measures analysis.
Changes in periperal blood platelets | Day 1-28
  Comparison of the course of plateletscounts at full blood counts among the treatment arm, as assessed by repeated measures analysis.
Changes in blood hemoglobin levels | Day 1-28
  Course of blood hemoglobin
Changes in blood creatinine levels | Day 1-28
  Course of blood creatine levels
Changes in blood albumin | Day 1-28
  Course of blood albumin levels
Changes in blood bilirubin | Day 1-28
  Course of blood bilirubin levles
Changes in blood LDH | Day 1-28
  Course of blood LDH levels
Changes in blood AST | Day 1-28
  Course of blood AST levels
Changes in blood ALT | Day 1-28
  Course of blood ALT levels
Changes in blood CK | Day 1-28
  Course of blood CK levels
Changes in blood C-reactive protein | Day 1-28
  Course of blood C-reactive protein levels
Changes in blood IL-6 | Day 1-28
  Course of blood IL-6 levels
Changes in blood protrombine time (INR) | Day 1-28
  Course of blood protrombine time (INR)
Changes in blood ferritin | Day 1-28
  Course of blood ferritin levels
Changes in blood troponin T | Day 1-28
  Course of blood troponin T levels
Changes in blood triglycerides | Day 1-28
  Course of blood triglycerides levels
Changes in blood HDL-colesterol | Day 1-28
  Course of blood HDL-colesterol levels
Changes in blood total colesterol | Day 1-28
  Course of blood total colesterol levels
Changes in blood D-Dimer | Day 1-28
  Course of blood D-Dimer levels
Changes in PaO2 at arterial gas analysis | Day 1-28
  Course of PaO2 at arterial gas analysis and PaO2/FiO2
Changes in PaO2/FiO2 | Day 1-28
  Course of PaO2/FiO2
Development of late complications | 6 months
  Death
Development of late complications | 6 months
  New Hospital admissions
Development of late complications | 6 months
  Proportion of patients developing new medical conditions in each interventional arm as compared to the control arm. Specific focus to:
  * new-onset interstitial lung disease
  * new onset respiratory failure requiring O2 therapy or ventilation therapy at home
  * thromboembolic event
  * ischemic events (stroke, acute coronary syndromes, pe-ripheral ischemias)
  * arterial hypertension
Development of late complications | 6 months
  Proportion of patients with FVC < 70% of predicted, FEV1 < 70% predicted and DLCO < 80% predicted

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Galli, MD, PhD, Principal Investigator — ASST Fatebenefratelli Sacco and Milan University
Locations (21):
- Italy (21):
  - Ospedali Riuniti delle Marche, Ancona
  - Ospedale Parini, Aosta
  - Ospedale SS Annunziata -Chieti, Chieti
  - Ospedale S Anna, Como
  - Ospedale di Ferrara, Ferrara
  - Ospedale di Firenze and Empoli, Florence
  - Ospedali Galliera, Genova
  - H Goretti, Latina
  - Ospedale Manzoni, Lecco
  - Ospedale di Legnago, Legnago
  - Ospedale di Legnano, Legnano
  - ASST Fatebenefratelli-Sacco, Milan
  - ASST Santi Paolo e Carlo, Milan
  - IRCCS San Raffaele, Milan
  - Ospedale di Perugia, Perugia
  - Ospedale San Salvatore, Pesaro
  - Ospedali di Prato e Pistoia, Prato
  - Policlinico Tor Vergata, Roma
  - Ospedale Cattinara e Maggiore, Trieste
  - Ospedale di Udine, Udine
  - Azienda Ospedaliera Integrata -Verona, Verona

IPD SHARING:
Plan to Share IPD: No
The e-CRF platform (Cloud-R) ensures data protection and satisties all quality requirements for data management and protection of patients confidentiality.
  Confidential data will be available only for physicians in charge of individual patients.
  Anonymized data will be made available to other research upon written request accompanied with a motivation and a scientific rationale